CLINICAL TRIAL: NCT04587869
Title: Still Climbin': A Randomized Controlled Trial to Improve Coping, Medical Mistrust, and Healthcare Engagement Among Black Sexual Minority Men
Brief Title: Still Climbin': An Intervention to Improve Coping Among Black Sexual Minority Men
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: NIH terminated the study due to shifted policy priorities
Sponsor: RAND (Other)
Collaborators: University of Massachusetts, Boston (Other); University of Southern California (Other); APLA Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01MD014722 (NIH)
Record Dates: First submitted 2020-10-01; First posted 2020-10-14 (Actual); Results first posted 2025-11-13 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-10

CONDITIONS: Discrimination, Social; Health Care Utilization
Keywords: Black/African American sexual minority men
MeSH Terms: conditions — Social Discrimination; Patient Acceptance of Health Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor does not randomize participant until after the baseline assessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention is an 8-session cognitive behavior therapy (CBT) group intervention that addresses coping with discrimination and medical mistrust among Black sexual minority men (SMM).
  Interventions: Behavioral: CBT Coping Intervention
- No-treatment control (No Intervention): Participants who are assigned to the control group will not receive the intervention.

INTERVENTIONS:
Behavioral: CBT Coping Intervention — A cognitive behavior therapy group intervention that addresses coping with discrimination and medical mistrust among Black sexual minority men (SMM).
  Arms: Intervention

SUMMARY:
This study consists of a randomized controlled trial of a multi-session cognitive behavior therapy (CBT) group intervention that addresses coping with discrimination and medical mistrust among Black sexual minority men (SMM). Primary intervention objectives include increasing health care engagement and receipt of evidence-based preventive care, as well as better coping and reduced anticipated and internalized stigma, and medical mistrust among intervention participants.

DETAILED DESCRIPTION:
This study is a randomized controlled trial of Still Climbin', an 8-session cognitive behavior therapy (CBT) group intervention that addresses coping with discrimination and medical mistrust among Black sexual minority men (SMM). Designed to be flexible for use in community settings, this intervention was developed in partnership with community stakeholders who emphasized the need for a community-based program outside of the health care system, and without a specific disease focus. It intends to give Black SMM a safe space to receive support for the whole of their identity and to openly discuss barriers to health care. Participants will be followed for 12 months. The effectiveness of the Still Climbin' intervention will be assessed on health care engagement and receipt of evidence-based preventive care, through surveys administered at multiple points throughout the intervention period. These outcomes will be confirmed with information from medical records. A total of 370 Black participants will be recruited and randomly assign 185 to receive the coping intervention and 185 to a no-treatment control. There will be about 10 groups of about 15 participants each for both intervention and control. Participants will be randomized to an intervention or control group after they complete the baseline survey. Participants will complete four surveys, starting with the baseline survey, and followed by 4-, 8-, and 12-month post-baseline follow-up surveys to assess health care engagement and receipt of evidence-based preventive care (e.g., cancer and diabetes screening, cardiovascular disease prevention, influenza vaccination, HIV prevention), and other topics such as coping strategies, stigma, and discrimination. The intervention is hypothesized to show increased health care engagement and receipt of evidence-based preventive care, in addition to better coping and reduced medical mistrust than the control group.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Biologically male at birth
* Identify as male
* Self-identify as a Black/African American
* Report having sex with men in the past 24 months
* Anticipate being available for the next 12 months to attend study visits
* Able to interact and communicate in written and spoken English.

Exclusion Criteria:

* Unwilling/Unable to provide informed consent
* Cisgender women
* Transgender women
* Transgender men

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Biologically male at birth; Identify as male
Enrollment: 369 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Bogart, PhD, Principal Investigator — RAND
Locations (1):
- APLA Health, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Following publication of the main study papers, de-identified survey data will be made publicly available to researchers who successfully complete a registration process after requesting to use the data. The data made available will not contain any direct or indirect identifiers. Users must agree to the conditions of use governing access to the public release data, including restrictions against attempting to identify study participants, destruction of the data after analyses are completed, reporting responsibilities, restrictions on redistribution of the data to third parties, and proper acknowledgement of the data resource.
Time Frame: For three years, following publication of the main study papers.
Access Criteria: Users must agree to the conditions of use governing access to the public release data, including restrictions against attempting to identify study participants, destruction of the data after analyses are completed, reporting responsibilities, restrictions on redistribution of the data to third parties, and proper acknowledgement of the data resource. Users must notify the institutional review board of their institution of their intention to use the data and their procedures for data management and security. Users must submit proposals regarding intended use of the data; the RAND study team and the RAND Human Subjects Protections Committee (HSPC) will determine the scientific soundness of the proposal as part of the decision for the researcher to be able to access the dataset.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | No-treatment Control
Started | 171 | 198
Completed | 125 | 137
Not Completed | 46 | 61
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 27 | 34
Not completed — Grant Termination | 13 | 25
Not completed — too busy | 2 | 0
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | No-treatment Control | Total
Number analyzed (Participants) | 171 | 198 | 369
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.73 (13.27) | 44.73 (12.37) | 44.73 (12.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 171 | 198 | 369
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 166 | 190 | 356
  White | 0 | 0 | 0
  More than one race | 5 | 8 | 13
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 171 | 198 | 369
Inadequate healthcare utilization [Count of Participants; unit: Participants] — Indicator that the individual reported (1) fewer than 1 ambulatory visit AND (2) at least 1 emergency department visit (without subsequent hospitalization), or at least 1 hospitalization in the past 4 months before baseline Population: This outcome was missing for 5 participants (1.4%) who did not respond to at least one of 3 items asking about hospital visits, ER visits, and urgent care visits
  Participants
    number analyzed (Participants) | 167 | 197 | 364
    (all) | 35 | 53 | 88
Proportion of evidence-based care components received [Mean (Standard Deviation); unit: proportion] — For each individual, this measure is the number of components that were received divided by the number of components they were eligible for, expressed as a proportion. 25 components were evaluated and eligibility for each component varies by individual.
  proportion | 0.59 (0.22) | 0.60 (0.22) | 0.60 (0.22)
Adaptive coping (social support seeking) [Mean (Standard Deviation); unit: units on a 4-point scale (range 1-4)] — Population: This outcome was missing for n=4 (1.1%), participants who did not respond to any of the 4 survey items included in this scale
  units on a 4-point scale (range 1-4)
    number analyzed (Participants) | 171 | 194 | 365
    (all) | 2.65 (0.91) | 2.57 (0.92) | 2.61 (0.92)

OUTCOME MEASURES:

1. Primary Outcome: Inadequate Healthcare Utilization
Description: Indicator that the individual reported (1) fewer than 1 ambulatory visit AND (2) at least 1 emergency department visit (without subsequent hospitalization) or at least 1 hospitalization in the past 4 months at any of the 3 follow-up assessments (4, 8, and 12 months post-baseline)
Time Frame: baseline to 12-month post-baseline
Population: The outcome is missing for all participants (n=53) who did not participate in any follow-up surveys (nonresponse weights were used to account for potential bias). The outcome was never missing among those who participated in any follow-up surveys.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | No-treatment Control
Number analyzed (Participants) | 148 | 168
Participants | 41 | 39
Statistical Analysis 1: Comparison: Intervention vs No-treatment Control; Nonresponse weights were employed to account for potential bias from excluding participants who did not complete any follow-up assessments; Test type: Superiority; p = .44, Regression, Logistic; Result was adjusted for HIV status and age (dichotomized at 50+ vs. <50), as those characteristics were used to stratify sampling; Odds Ratio (OR) = 1.23, 95% CI 2-sided [.73 to 2.07] — Result is for indicator of assignment to intervention arm (vs. control)

2. Primary Outcome: Proportion of Evidence-based Care Components Received Across Follow-up Assessments
Description: For each individual, this measure is the number of components that were received at any time across the 3 follow-up assessments divided by the number of components they were eligible for at any time across the 3 follow-up assessments, expressed as a proportion. 25 components were evaluated and eligibility for each component varies by individual and follow-up period.
Time Frame: baseline to 12 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: proportion
Arm/Group | Intervention | No-treatment Control
Number analyzed (Participants) | 148 | 168
proportion | .46 (.22) | .47 (.23)
Statistical Analysis 1: Comparison: Intervention vs No-treatment Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .47, Regression, Linear; [statistical method as in outcome 1, analysis 1]; Slope = -0.02, Standard Error of Mean 0.02 — Result is for indicator of assignment to intervention arm (vs. control)

3. Secondary Outcome: Adaptive Coping Strategies (Social Support Seeking)
Description: Average adaptive coping rating on the Brief COPE scale, social support items (higher=better coping; range=1-4)
Time Frame: 4-, 8-, and 12-months post-baseline
Population: The outcome is missing for all participants (n=53) who did not participate in any follow-up surveys. The outcome is missing for an additional n=10 (3.2%) participants who did not complete any of the 4 survey items included in the scale.
  Because this measure was analyzed in a repeated measures regression framework where each participant may contribute up to 3 observations (and may or may not complete each assessment), the sample size varies by assessment.
Measure: Mean (Standard Deviation); unit: units on a scale (range 1-4)
Arm/Group | Intervention | No-treatment Control
Number analyzed (Participants) | 143 | 163
units on a scale (range 1-4)
  4-month assessment: number analyzed (Participants) | 119 | 137
  4-month assessment | 2.60 (0.96) | 2.50 (0.96)
  8-month assessment: number analyzed (Participants) | 114 | 126
  8-month assessment | 2.77 (0.96) | 2.56 (0.92)
  12-month assessment: number analyzed (Participants) | 120 | 134
  12-month assessment | 2.61 (0.92) | 2.41 (0.91)
Statistical Analysis 1: Comparison: Intervention vs No-treatment Control; Unlike the two primary outcomes which have a single value for each participant, for this outcome we employed a repeated measures style structure with one record for each of up to 3 FU observations. A sandwich estimator (SAS Proc Surveyreg) was employed to account for clustering of observations within participant. In addition, nonresponse weights were employed to account for potential bias from excluding participants who did not complete any follow-up assessments; Test type: Superiority; p = .02, Regression, Linear; [statistical method as in outcome 1, analysis 1]; Slope = 0.19, Standard Error of Mean 0.08 — Slope is adjusted regression coefficient for indicator of intervention arm (so mean of outcome across follow-ups was 0.19 higher for intervention vs. control)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Intervention | No-treatment Control
All-Cause Mortality (participants affected / at risk) | 1/171 | 0/198
Serious Adverse Events (participants affected / at risk) | 22/171 | 17/198
Other Adverse Events (participants affected / at risk) | 0/171 | 0/198
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=171) | No-treatment Control (N=198)
Stroke and other nervous system disorder (Nervous system disorders) | 6 (6) | 2 (2)
Cardiac-related hospitalization (Cardiac disorders) | 5 (5) | 3 (3)
GI related hospitalization (Gastrointestinal disorders) | 1 (1) | 1 (1)
Respiratory related hospitalization (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Infection - hospitalization (Infections and infestations) | 2 (2) | 1 (1)
Accidents (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
General -surgery due to pre-existing conditions (Surgical and medical procedures) | 1 (1) | 4 (4)
Kidney failure (Renal and urinary disorders) | 0 (0) | 1 (1)
General hospitalization (Surgical and medical procedures) | 1 (1) | 0 (0) — reason unknown

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-01-13): https://cdn.clinicaltrials.gov/large-docs/69/NCT04587869/Prot_SAP_000.pdf
  • Informed Consent Form (2023-04-04): https://cdn.clinicaltrials.gov/large-docs/69/NCT04587869/ICF_001.pdf